CLINICAL TRIAL: NCT06434454
Title: EFT and Sleep Quality
Acronym: EFT STUDENT
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Bezmialem Vakif University (Other)
Responsible Party: Principal Investigator, Merve Meşedüzü, LECTURER, Bezmialem Vakif University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: E-54022451-050.04-137924; MMeseduzu (Other: BezmialemVU)
Record Dates: First submitted 2024-05-20; First posted 2024-05-30 (Actual); Last update posted 2024-05-30 (Actual); Status verified 2024-05

CONDITIONS: Sleep Quality
Keywords: student; sleep qualıty; emotioanal freedom techniques
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Intervention Model Description: The young individuals in the control group will be informed about the study, including its purpose and methodology, and their consent will be obtained. The control group will receive sleep education, consisting of two educational presentations provided 15 days apart. The questionnaires of the scales used for analysis will be administered to assess their sleep problems. The content of the education will be prepared based on the literature and will be reviewed by at least three experts.
  The young individuals in the experimental group will be informed about the study, including its purpose and methodology, and their consent will be obtained. Emotional Freedom Techniques (EFT) will be applied to groups of 20 individuals to improve sleep quality, and all scales will be administered beforehand. EFT will be applied twice, with a 15-day interval between sessions, and the same scale questionnaires will be administered again after the second EFT session. Subsequently, the analysis
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EXPERİMENTAL: EFT GROUP (Experimental): The young individuals in the intervention group will be informed about the study, including its purpose and methodology, and their consent will be obtained. Emotional Freedom Techniques (EFT) will be applied to groups of 20 individuals to improve sleep quality, and all scales will be administered beforehand. EFT will be applied twice, with a 15-day interval between sessions, and the same scale questionnaires will be administered again after the second EFT session. Subsequently, the analysis will be conducted.
  Interventions: Behavioral: EFT Group:Emotional Free Technıcal
- CONTROL GROUP (No Intervention): The young individuals in the control group will be informed about the study, including its purpose and methodology, and their consent will be obtained. The control group will receive sleep education, consisting of two educational presentations provided 15 days apart. The questionnaires of the scales used for analysis will be administered to assess their sleep problems. The content of the education will be prepared based on the literature and will be reviewed by at least three experts.

INTERVENTIONS:
Behavioral: EFT Group:Emotional Free Technıcal — The young individuals in the intervention group will be informed about the study, including its purpose and methodology, and their consent will be obtained. Emotional Freedom Techniques (EFT) will be applied to groups of 20 individuals to improve sleep quality, and all scales will be administered beforehand. EFT will be applied twice, with a 15-day interval between sessions, and the same scale questionnaires will be administered again after the second EFT session. Subsequently, the analysis will be conducted.
  Other Names: emotional free technıcal
  Arms: EXPERİMENTAL: EFT GROUP

SUMMARY:
The purpose of this clinical study is to determine whether the application of EFT (Emotional Freedom Techniques) is effective in reducing sleep problems among university students. Additionally, the study aims to gather information on the safety of EFT application. The primary questions it seeks to answer are:

Does EFT application reduce sleep problems among university students? Is EFT application feasible for addressing sleep problems in university students? Researchers will compare the effectiveness of EFT to traditional sleep education on non-pharmacological interventions for preventing sleep problems among university students.

Participants:

Pre-EFT application survey scale questions will be asked to university students.

EFT will be applied once by the researcher to university students. EFT will be applied a second time by the researcher to university students 15 days after the initial application.

For control, the same survey scale questions will be asked to the same students one day after the EFT application for post-test purposes.

The same procedures will be applied in the same manner to the control group that will receive education.

DETAILED DESCRIPTION:
DATA COLLECTION TOOLS AND THEIR FEATURES For data collection, a questionnaire including socio-demographic characteristics, the Insomnia Severity Index, the Epworth Sleepiness Scale, and the Pittsburgh Sleep Quality Index will be used.

1. Personal Information Form The personal information form, prepared by the researchers, includes questions about socio-demographic characteristics such as age and gender. The last part of the questionnaire consists of questions evaluating the sleep status of the participants.
2. Insomnia Severity Index (ISI) This scale, developed to determine the severity of insomnia symptoms, can be used in both general population screenings and clinical assessments of insomnia. It is a seven-item, five-point Likert-type scale. Each item is scored between 0 and 4, with the total score ranging from 0 to 28. Scores of 0-7 indicate no clinically significant insomnia, 8-14 indicate subthreshold insomnia, 15-21 indicate clinical insomnia (moderate severity), and 22-28 indicate severe clinical insomnia.
3. Epworth Sleepiness Scale (ESS) The ESS is an easy-to-administer and widely used scale. It is a four-point Likert-type scale. Each item is scored 0, 1, 2, or 3, with higher scores indicating greater daytime sleepiness. It aims to measure the general level of daytime sleepiness and is a simple self-report tool.
4. Pittsburgh Sleep Quality Index (PSQI) The PSQI& index comprises 18 items grouped into 7 component scores. Each item is evaluated on a scale of 3 points. The sum of the seven component scores provides the total PSQI score, ranging from 0 to 21. Higher total scores indicate poorer sleep quality. A total PSQI score of 0-4 signifies good sleep quality, while scores between 5-21 indicate poor sleep quality.

   indicates and shows a serious deterioration in at least two components or moderate deterioration in three components of the PSQI.
5. Fatigue Severity Scale (FSS) The FSS consists of 9 questions measuring the degree of fatigue experienced in the past week. Each question is rated on a scale from 0 (strongly disagree) to 7 (strongly agree), and the total score is the sum of these ratings. The highest possible total score is 63. A score of 36 or above indicates significant fatigue.
6. Sleep Education (control group):

The sleep education content will be prepared by the researcher based on the literature and will be reviewed by at least three experts.

ELIGIBILITY:
* Inclusion Criteria:

  * Görsel Analog Ölçeğe (VAS) göre 5 ve üzerinde uyku sorunu bildiren öğrenciler
  * 18-24 yaş aralığında olan öğrenciler
  * Herhangi bir kronik hastalığı bulunmayan öğrenciler
  * Araştırmaya gönüllü olarak katılmak isteyen öğrenciler yer almaktadır.
* Exclusion Criteria:

  * Individuals who wish to withdraw from the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 74 (Estimated)
Dates: Start 2024-06-20 (Estimated); Primary Completion 2024-08-20 (Estimated); Study Completion 2024-09-20 (Estimated)

PRIMARY OUTCOMES:
Insomnia Severity Index Scale | 1 months
  This scale is a seven-item, five-point Likert-type scale. Each item is scored between 0 and 4, with the total score ranging from 0 to 28. Scores of 0-7 indicate no clinically significant insomnia, 8-14 indicate subthreshold insomnia, 15-21 indicate clinical insomnia (moderate severity), and 22-28 indicate severe clinical insomnia

SECONDARY OUTCOMES:
Epworth Sleepiness Scale (ESS) | 1 months
  The ESS is a four-point Likert-type scale. Each item is scored 0, 1, 2, or 3, with higher scores indicating greater daytime sleepiness. It aims to measure the general level of daytime sleepiness and is a simple self-report tool.

OTHER OUTCOMES:
Fatigue Severity Scale (FSS) | one month
  The FSS consists of 9 questions measuring the degree of fatigue experienced in the past week. Each question is rated on a scale from 0 (strongly disagree) to 7 (strongly agree), and the total score is the sum of these ratings. The highest possible total score is 63. A score of 36 or above indicates significant fatigue.
Pittsburgh Sleep Quality Index (PSQI) | one month
  The index comprises 18 items grouped into 7 component scores. Each item is evaluated on a scale of 3 points. The sum of the seven component scores provides the total PSQI score, ranging from 0 to 21. Higher total scores indicate poorer sleep quality. A total PSQI score of 0-4 signifies good sleep quality, while scores between 5-21 indicate poor sleep quality. indicates and shows a serious deterioration in at least two components or moderate deterioration in three components of the PSQI.

CONTACTS AND LOCATIONS:
Locations (1):
- Bezmialem Vakif Universty, Istanbul, Topkapı Mahallesi, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided